CLINICAL TRIAL: NCT01362920
Title: Diagnostic and Prognostic Value of Serial PCT Measurements in Critically Ill Patients
Brief Title: Diagnostic and Prognostic Value of Serial Procalcitonin (PCT) Measurements in Critically Ill Patients
Acronym: PCT
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor
Other Study IDs: PCT-001
Record Dates: First submitted 2011-04-06; First posted 2011-06-01 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Sepsis
Keywords: Sepsis; Septic shock; Procalcitonin; PCT
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sepsis or Septic shock cohort
- Non-sepsis or non-Septic shock cohort

SUMMARY:
In 2005, the Food and Drug Administration (FDA) approved procalcitonin in conjunction with other laboratory markers to aid in the risk assessment of critically ill patients with severe infection (sepsis). Although considerable literature exists regarding the usefulness of Procalcitonin (PCT) as a marker of sepsis, there are still potential uses for PCT measurements that are not yet explored and its value among the critically ill patients remains unclear. This study seeks to better understand the usefulness of measuring PCT values in patients admitted to the Medical ICU for a variety of reasons and in particular with severe infection (sepsis).

DETAILED DESCRIPTION:
Procalcitonin (PCT) is a 116 amino acid peptide that has an approximate MW of 14.5 kDa and belongs to the calcitonin (CT) superfamily of peptides. Transcription of the CALC-1 gene for PCT is usually suppressed in the non-neuroendocrine tissue, except in the C cells of the thyroid gland where its expression produces PCT, the precursor of CT in healthy individuals and in the absence of infection.

In the presence of microbial infection, circulating levels of calcitonin precursors (CTpr), including PCT, increase up to several thousand-fold.1 In addition to being a marker of microbial infection, PCT also acts as a modulator of the host inflammatory reaction. In an animal model of sepsis, administration of exogenous human PCT worsened outcome, whereas neutralization of endogenous PCT improved survival.

There are several inflammatory laboratory markers, like tumor necrosis factor (TNF)-α, interleukin (IL)-1, IL-6 and C-reactive protein (CRP), but they are non- specific for infection and can be caused by conditions like pancreatitis, burns, trauma or acute lung injury. The non-specific nature of clinical and laboratory parameters for microbial infection makes it difficult to evaluate patients with potential infection. In addition to the lack of specificity, traditional laboratory and clinical indicators of sepsis are not temporally concordant with the course of illness. As a result, these tests are not reliable to evaluate the response to therapeutic interventions in real time.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients admitted to the Medical Intensive Care Unit of the Cleveland Clinic with an anticipated MICU stay of ≥ 12hrs

Exclusion Criteria:

* Age less than 18-years of age and/or an expected MICU stay of less than 12-hrs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prospective-observational study design in which a PCT measurement will be obtained on admission to the Medical Intensive Care Unit (MICU) and then daily (as clinically available)until discharge from the unit or death.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Development of organ failure | Current hospitalization (participants will be followed for the duration of hospital stay; an expected average of 7-days)
Development and resolution of shock using a cut-off PCT of >0.5ng/mL | ICU stay (participants will be followed for the duration of hospital stay; an expected average of 7-days)
ICU and Hospital Mortality | current hospitalization or 28-day post ICU admission for ICU survivors

SECONDARY OUTCOMES:
Development of hospital acquired infections (catheter related blood stream infection, development of multidrug resistant infections, ventilator associated pneumonia) | Current hospitalization (participants will be followed for the duration of hospital stay; an expected average of 7-days)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge A Guzman, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States